CLINICAL TRIAL: NCT06068608
Title: A Randomized, Double-blind, Placebo-Controlled, Single Ascending Dose, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TNM005 and to Characterize the Pharmacodynamics of TNM005 and VARIZIG in Healthy Adult Volunteers
Brief Title: A Trial to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic Profile of TNM005 in Healthy Adult Subjectsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TNM005-101
Record Dates: First submitted 2023-09-16; First posted 2023-10-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2023-09

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — varicella-zoster immune globulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TNM005 dose level 1/placebo (Experimental): TNM005 on dose level 1 /placebo
  Interventions: Drug: TNM005; Drug: Placebo
- TNM005 dose level 2/placebo (Experimental): TNM005 on different dose level 2 /placebo
  Interventions: Drug: TNM005; Drug: Placebo
- TNM005 level 3/placebo (Experimental): TNM005 on dose level 3 /placebo
  Interventions: Drug: TNM005; Drug: Placebo
- TNM005 dose level 4/placebo (Experimental): TNM005 on dose level 4 /placebo
  Interventions: Drug: TNM005; Drug: Placebo
- TNM005 dose level 5/placebo (Experimental): TNM005 on dose level 5 /placebo
  Interventions: Drug: TNM005; Drug: Placebo
- VARIZIG (Active Comparator): VARIZIG 625 IU
  Interventions: Drug: VariZIG

INTERVENTIONS:
Drug: TNM005 — single,intramuscular injection
  Arms: TNM005 dose level 1/placebo; TNM005 dose level 2/placebo; TNM005 dose level 4/placebo; TNM005 dose level 5/placebo; TNM005 level 3/placebo
Drug: Placebo — single,intramuscular injection
  Arms: TNM005 dose level 1/placebo; TNM005 dose level 2/placebo; TNM005 dose level 4/placebo; TNM005 dose level 5/placebo; TNM005 level 3/placebo
Drug: VariZIG — a single dose of VARIZIG 625 IU,intramuscular injection
  Arms: VARIZIG

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of TNM005 following a single dose by intramuscular (IM) administration in healthy adult subjects The main questions it aims to answer are:1. safety profile；2. PK properties 3. PD properties

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose, phase 1 study designed to evaluate the safety, tolerability, PK, PD (anti-VZV antibody level), and immunogenicity of TNM005, as well as to characterize the PD of VARIZIG, in healthy adult volunteers.

The study also includes a cohort in which eight subjects will receive a single dose of VARIZIG 625 IU. This cohort will be conducted in an open-label fashion and may be initiated as early as the first TNM005 cohort is dosed.

The study include periods of Screening (up to 28 days), in-patient (treatment on Day 1), and safety follow-up until Day 120.

ELIGIBILITY:
Inclusion Criteria:

* 1) Signed and dated written informed consent;
* 2) Are willing and able to comply with scheduled visits, blood sampling, laboratory tests, and other study procedures;
* 3) Healthy males or females, 18-55 years of age (both inclusive);
* 4) Body mass index (BMI) within 18.5-31.0 kg/m2 (both inclusive) and body weight ≥50.0 kg for males and ≥45.0 kg for females;
* 5) Have no clinically significant abnormality on physical examination, vital signs, 12-lead ECG, and clinical laboratory tests as determined by the Investigator;
* 6) Females must be either surgically sterile or under post-menopausal status at Screening or agree to use a highly effective method of contraception from screening until 120 days after IMP dosing. In addition, males who are sexually active and partners of women of childbearing potential must agree to use effective contraception from screening until 120 days after drug administration.

Exclusion Criteria:

* 1) History or evidence of any other acute or chronic disease that, in the opinion of the Investigator, may interfere with the evaluation of the safety or immunogenicity of the drug or compromise the safety of the subject;
* 2) History of surgery (except minor outpatient surgery) within three months prior to screening or planned surgery during the study;
* 3) History of receiving monoclonal antibody, immunoglobulin, or blood products within six months prior to dosing;
* 4) Receipt of systemic immunosuppressive medications;
* 5) Exposure to any live attenuated vaccine within four weeks prior to drug administration;
* 6) History of receiving vaccine(s) against zoster;
* 7) Use of any other drug, including over-the-counter medications, and herbs, within 14 days prior to the drug administration or five half-lives of the drug, whichever is longer, except for contraceptive medication in women of childbearing potential (WOCBP), or concomitant medications that are considered necessary for the subject's welfare and unlikely to interfere with the study;
* 8) Donated blood >400 mL or significant blood loss equivalent to 400 mL within one month before Screening; or plasma donation within 14 days before Screening; or any plan of blood or blood product donation during the study;
* 9) Positive test at a screening of any of the following: hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibody, or human immunodeficiency virus (HIV) antigen/antibody;
* 10) Known or suspected history of drug abuse within the past five years or with a positive urine drug test at Screening or on Day -1;
* 11) History of significant alcohol abuse within six months prior to screening or any indication of regular use of more than 14 units of alcohol per week or taking a product containing alcohol two days prior to dosing, or having a positive alcohol breath test on Day -1;
* 12) Use of ≥five cigarettes or equivalent nicotine-containing product per day on average over three months prior to Screening; or unwilling to refrain from nicotine products during study participation;
* 13) History of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG-fusion protein;
* 14) History of allergic or anaphylactic reaction to blood products (only for VARIZIG cohort);
* 15) IgA deficient subjects at risk for hypersensitivity reaction (only for VARIZIG cohort);
* 16) Subjects at high risk for thrombotic events, including those with a history of venous or arterial thrombosis, atherosclerosis, or multiple cardiovascular risk factors (only for VARIZIG cohort);
* 17) Participation in any other clinical studies with chemical or biological drugs or devices within four weeks or five times the half-life of the specific drug/biologics (whichever is longer) before drug administration;
* 18) Nursing mothers or pregnant women;
* 19) Subjects considered unsuitable for participating in the study in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | Up to 120 days post dosing
Number of participants Physical examinations abnormalities | Up to 120 days post dosing
  Physical examination includes assessments of general appearance, skin, lymph nodes, head.neck, lung, heart, abdomen, spine, extremities, nervous system, etc.
Number of participants with abnormalities of vital signs | Up to 120 days post dosing
  Vital signs measured include blood pressure, pulse rate, temperature, and respiration rate.
Number of participants with abnormalities of 12-lead electrocardiogram (ECG) parameters | Up to 120 days post dosing
  ECG parameters include heart rate, PR interval, RR interval, ORS duration, QTcF interval.
Number of participants with abnormalities of clinical laboratory tests | Up to 120 days post dosing
  Clinical laboratory tests include hematology, biochemistry, coagulation, and urinalysis.

SECONDARY OUTCOMES:
AUC0-t | Up to 120 days post dosing
  Area under the plasma concentration-time curve from time 0 (predose) to the last time point with a detectable plasma concentration (Tlast.).
AUC0-∞ | Up to 120 days post dosing
  Area under the plasma concentration-time curve from time 0 (predose) extrapolated to infinite time.
Cmax | Up to 120days post dosing
  Maximum plasma concentration
Tmax | Up to 120 days post dosing
  Time to reach maximum plasma concentration
t1/2 | Up to 120days post dosing
  Elimination half-life
λz | Up to 120days post dosing
  Terminal disposition rate constant
CL/F | Up to 120days post dosing
  Apparent clearance
Vd/F | Up to 120days post dosing
  Apparent volume of distribution
t1/2 of anti-varicella-zoster virus (VZV) antibody level (both baseline corrected and uncorrected) | Up to 120days post dosing
  Elimination half-life of antibody level of anti-VZV
ADA | Up to 120days post dosing
  Incidence of anti-drug antibody (ADA) to TNM005 in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ahad Sabet, MD, Principal Investigator — ICON plc
Locations (1):
- ICON, plc, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No